CLINICAL TRIAL: NCT06068660
Title: Effects of a Goal-Oriented Care on Health Outcome in Patients With Unplanned Dialysis After Discharge
Brief Title: Effects of a Goal-Oriented Care Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202101313A3
Record Dates: First submitted 2023-09-20; First posted 2023-10-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases; Acute on Chronic Renal Failure; Acute Kidney Injury
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): The experimental group during hospitalization additionally received 40 minutes of one-on-one education three times a week for three weeks, as the Goal-Oriented Care program for 6 hours in total, followed by telephone sessions of 20 minutes every month for six months post-discharge.
  Interventions: Behavioral: The Goal-Oriented Care program; Behavioral: The routine health education
- The control group (Active Comparator): The control group received routine health education
  Interventions: Behavioral: The routine health education

INTERVENTIONS:
Behavioral: The Goal-Oriented Care program — The Goal-Oriented Care Interventions The GOC intervention included the following steps: respecting the participant's values in setting goals, considering direct and indirect factors influencing the goals, communicating and setting goals, implementing goal-oriented strategies, and evaluating goals while adjusting the content of the strategies.
  Arms: The experimental group
Behavioral: The routine health education — The control group received routine education, which consisted of oral education and provision of educational pamphlets by nurses during hospitalization.

SUMMARY:
This study was a clinical trial. This study aimed to evaluate the effects of Goal-Oriented Care intervention on blood pressure, percentage of interdialytic weight gain, self-management behaviors, and quality of life in hospitalized patients with unplanned dialysis at three and six-months post-discharge. This study was an experimental design in a medical center in Southern Taiwan. A cluster sample method was selected for each two wards from four nephrology wards and was randomly assigned to the experimental and control groups. The enrolled patients were assigned to the experimental and control groups according to different wards' admission. The inclusion criteria were: (1) patients who received unplanned dialysis during hospitalization; (2) aged between 20 and 80 years; (3) not undergoing renal replacement therapy before recruitment; (4) alert consciousness status and ability to communicate; (5) ability to perform self-management behaviors. The exclusion criteria were a history of psychiatric illness, any active infection and inability to communicate or understand the educational process. Each group consisted of 46 participants. Both groups received routine health education. However, the experimental group during hospitalization additionally received 40 minutes of one-on-one education three times a week for three weeks, as the Goal-Oriented Care program for 6 hours in total, followed by telephone sessions of 20 minutes every month for six months post-discharge. On receiving the third dialysis, baseline data including self-report questionnaires assessed participants' demographic and disease characteristics and medical record reports for blood pressure and percentage of interdialytic weight gain were collected. A week after discharge, self-management behaviors and quality of life baseline data were assessed using self-reported questionnaires and these were followed up at three and six-months post-discharge, which then also included blood pressure and percentage of interdialytic weight gain.Generalized estimating equations were used to assess changes amounts in each outcome variable from the baseline to three months and six-months post-discharge between two groups.

DETAILED DESCRIPTION:
On receiving the third dialysis, baseline data including self-report questionnaires assessed participants' demographic and disease characteristics and medical record reports for blood pressure and percentage of interdialytic weight gain were collected. A week after discharge, self-management behaviors and quality of life baseline data were assessed using self-reported questionnaires and these were followed up at three and six-months post-discharge, which then also included blood pressure and percentage of interdialytic weight gain. All data were analyzed using the computer-based statistical software package SPSS, version 20.0. Descriptive statistics were calculated to examine the distribution of the study variables as mean, standard deviation and percentage among participants. Inferential statistics included the chi-square test, independent two-sample t-test, and paired sample t-test. Generalized estimating equations were used to assess changes amounts in each outcome variable from the baseline to three months and six-months post-discharge between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. patients who received unplanned dialysis during hospitalization;
2. aged between 20 and 80 years;
3. not undergoing renal replacement therapy before recruitment;
4. alert consciousness status and ability to communicate;
5. ability to perform self-management behaviors.

Exclusion Criteria:

The exclusion criteria were a history of psychiatric illness, any active infection and inability to communicate or understand the educational process.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurements | Baseline measurements were taken in a supine position during the third hemodialysis session and recorded systolic and diastolic blood pressures. Follow-up measurements were taken before each hemodialysis session at three and six months after discharge.
  Blood pressure measurements were performed by dialysis technicians using regularly maintained blood pressure monitors.
Percentage of interdialytic weight gain (IDWG%) during dialysis | The average of all measurements taken during the two weeks after the third dialysis session served as the baseline, while the average of all measurements taken every three months during the three- and six-month follow-up periods was recorded.
  Interdialytic weight gain percentage (IDWG%) was calculated as the difference between the weight at the start of dialysis and the weight after the previous dialysis session, divided by the dry weight set by the physician, expressed as a percentage.
The hemodialysis self-management scale 20 items and measures the execution of problem-solving, emotional management, self-care, and partner relationships | Baseline data collected from participants during their hospitalization after the third hemodialysis session. Follow-up data on self-management behaviors, and quality of life questionnaires were collected at three months and six months after discharge.
  The self-administered Chinese version of the Hemodialysis Self-Management Scale, developed by Song and Lin (Song & Lin 2009), was used. It consists of 20 items and measures the execution of problem-solving, emotional management, self-care, and partner relationships in the daily lives of dialysis patients. Responses were rated on a Likert scale ranging from "never" (scored as 1) to "always" (scored as 4). The total score ranges from 20 to 80, with higher scores indicating better self-management levels.
The physical component summary (PCS) and mental component summary (MCS) Quality of Life | Baseline data collected from participants during their hospitalization after the third hemodialysis session. Follow-up data on self-management behaviors, and quality of life questionnaires were collected at three months and six months after discharge.
  The Taiwan version of the 36-item Medical Outcome Study Short Form Health Survey (SF-36), translated by Lu et al. in 2003, was used to assess patients' physical and mental health-related quality of life within the past 30 days. The physical component summary (PCS) includes measurements of bodily functioning, physical role, pain, and general health. The mental component summary (MCS) includes measurements of vitality, emotional role, social functioning, and mental health. Scores were obtained through questionnaire responses and converted based on the SF-36 manual, with scores ranging from 0 to 100. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, Principal Investigator — Institutional Review Board Chang Gung Medical Foundation
Locations (1):
- ChangGungMH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No